CLINICAL TRIAL: NCT02043938
Title: 'Study of the Cerebral Effects of Sevoflurane, Propofol and Remifentanil as Measured by the Spontaneous Electro-encephalogram'
Brief Title: Improving Information Extraction From EEG on Cerebral Anesthetic Drug Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STRU0002
Record Dates: First submitted 2014-01-09; First posted 2014-01-23 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-03

CONDITIONS: Anesthesia
Keywords: Electroencephalography; pharmacological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Healthy Volunteers (Experimental): All healthy volunteers will receive four sessions of anesthesia with different common drug combinations while having SedLine EEG sensors placed on their forehead during these sessions to study the effects of these drugs on the brain. The sessions were: propofol (P), sevoflurane (S), propofol with remifentanil (PR), and sevoflurane with remifentanil (SR).
  Interventions: Device: SedLine EEG sensor

INTERVENTIONS:
Device: SedLine EEG sensor — Test subjects in each group will receive the same device intervention (SedLine EEG) to monitor their EEG waves.

SUMMARY:
This is an interventional, randomized controlled study in health volunteers that involves collecting data on raw EEG waves measuring various combinations of anesthetic drugs during standardized drug titration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 70 years
* Concerning the cognitive function: Volunteers are considered to have sufficient cognitive reserve if they are able to read and comprehend the patient information form, if they can adequately answer the anamnestic questions during the screening process and if they are allowed to provide legitimate written informed consent
* No selection will be made regarding ethnic background.
* For this study no control group has been selected as EEG is compared between episodes rather than between individuals (each volunteer is his/her own control)

Exclusion Criteria:

Volunteer refusal

* Volunteer < 18 years and >70 years
* Pregnancy
* Exclusion criteria are weight less than 70% or more than 130% of ideal body weight
* Neurological disorder (epilepsy, the presence of a brain tumor, a history of brain surgery, hydrocephalic disorders, depression needing treatment with anti-depressive drugs, a history of brain trauma, a subarachnoidal bleeding, TIA or cerebral infarct, psychosis or dementia , schizophrenia, alcohol or drug abuse).
* Diseases involving the cardiovascular system (hypertension, coronary artery disease, prior acute myocardial infarction, any valvular and/or myocardial disease involving decrease in ejection fraction, arrhythmias, which are either symptomatic or require continuous medication/pacemaker/automatic internal cardioverter defibrillator
* Pulmonary Diseases
* Gastric Diseases
* Endocrinologic diseases
* Recent use of psycho-active medication (benzodiazepines, anti-epileptic drugs, parkinson medication, anti-depressant drugs, opioids) or more than 20g of alcohol daily

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2015-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su H, Koomen JV, Eleveld DJ, Struys MMRF, Colin PJ. Pharmacodynamic mechanism-based interaction model for the haemodynamic effects of remifentanil and propofol in healthy volunteers. Br J Anaesth. 2023 Aug;131(2):222-233. doi: 10.1016/j.bja.2023.04.043. Epub 2023 Jun 22. PMID 37355412
- [Derived] Su H, Eleveld DJ, Struys MMRF, Colin PJ. Mechanism-based pharmacodynamic model for propofol haemodynamic effects in healthy volunteers☆. Br J Anaesth. 2022 May;128(5):806-816. doi: 10.1016/j.bja.2022.01.022. Epub 2022 Mar 3. PMID 35249706
- [Derived] Ramaswamy SM, Kuizenga MH, Weerink MAS, Vereecke HEM, Struys MMRF, Belur Nagaraj S. Frontal electroencephalogram based drug, sex, and age independent sedation level prediction using non-linear machine learning algorithms. J Clin Monit Comput. 2022 Feb;36(1):121-130. doi: 10.1007/s10877-020-00627-3. Epub 2020 Dec 14. PMID 33315176
- [Derived] Ramaswamy SM, Kuizenga MH, Weerink MAS, Vereecke HEM, Struys MMRF, Nagaraj SB. Novel drug-independent sedation level estimation based on machine learning of quantitative frontal electroencephalogram features in healthy volunteers. Br J Anaesth. 2019 Oct;123(4):479-487. doi: 10.1016/j.bja.2019.06.004. Epub 2019 Jul 18. PMID 31326088
- [Derived] Kuizenga MH, Colin PJ, Reyntjens KMEM, Touw DJ, Nalbat H, Knotnerus FH, Vereecke HEM, Struys MMRF. Test of neural inertia in humans during general anaesthesia. Br J Anaesth. 2018 Mar;120(3):525-536. doi: 10.1016/j.bja.2017.11.072. Epub 2017 Dec 1. PMID 29452809

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Thirty-six healthy volunteers received four sessions of anesthesia with different common drug combinations while having SedLine EEG sensors placed on their forehead during these sessions to study the effects of these drugs on the brain. The sessions were: propofol (P), sevoflurane (S), propofol with remifentanil (PR), and sevoflurane with remifentanil (SR).
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 46
Completed | 36
Not Completed | 10
Not completed — Withdrawal by Subject | 7
Not completed — Unable to place EEG sensors on patient | 1
Not completed — No show by subject | 1
Not completed — Investigator decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 43.3 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 36

OUTCOME MEASURES:

1. Primary Outcome: Patient State Index (PSI) Comparison, Baseline and Emax
Description: Patient State Index (PSI-1) is a processed EEG parameter that quantifies the level of EEG inhibition. A new algorithm (PSI-2) has been created to improve performance in low power EEG. PSI is unitless. It ranges between 100 and 0 (100 representing 'awake state', 0 denoting 'no detectable electrical brain activity'). PSI-1 and PSI-2 were compared in their correlation with measured propofol and sevoflurane concentrations with or without remifentanil (0, 2 ,or 4 ng/mL) via several estimated PD model parameters. In the data table, BL (Baseline) denotes PSI-2 measurements when no drug is present; Emax denotes PSI in the presence of the maximum drug effect; C50 is the drug concentration which produces 50% of the maximal drug effect (ug/mL for Propofol C50, vol% for Sevoflurane C50).
Time Frame: 6 weeks
Population: All 36 participants experienced all four interventions: Propofol only (P), Sevoflurane only (S), Propofol with Remifentanil (PR), and Sevoflurane with Remifentanil (SR).
Measure: Mean (Standard Error); unit: index
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
index
  No Drugs, PSI-2 (BL) | 85.1 (0.8)
  P, PSI-2 (Emax) | 63.1 (1.9)
  PR, PSI-2 (Emax) | 63.1 (1.9)
  S, PSI-2 (Emax) | 67.2 (2.3)
  SR, PSI-2 (Emax) | 67.2 (2.3)
  No Drugs, PSI-1 (BL) | 85.1 (0.8)
  P, PSI-1 (Emax) | 63.1 (1.9)
  PR, PSI-1 (Emax) | 63.1 (1.9)
  S, PSI-1 (Emax) | 0.152 (17.1)
  SR, PSI-1 (Emax) | 0.152 (17.1)

2. Other Pre Specified Outcome: Patient State Index (PSI) Comparison, C50 (Sevoflurane, Sevoflurane+Remifentanil)
Description: as for outcome 1
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: %vol
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
%vol
  S, PSI-2 (C50) | 1.22 (3.1)
  SR, PSI-2 (C50) | 1.22 (3.1)
  S, PSI-1 (C50) | 1.22 (3.1)
  SR, PSI-1 (C50) | 1.22 (3.1)

3. Other Pre Specified Outcome: Patient State Index (PSI) Comparison, C50 (Propofol, Propofol+Remifentanil)
Description: as for outcome 1
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
ug/mL
  P, PSI-2 (C50) | 1.63 (3.7)
  PR, PSI-2 (C50) | 1.63 (3.7)
  P, PSI-1 (C50) | 1.63 (3.7)
  PR, PSI-1 (C50) | 1.63 (3.7)

4. Other Pre Specified Outcome: Propofol, Sevoflurane, and Remifentanil Interaction.
Description: For all study groups (i.e. P, S, PR, and SR), the estimated PD model parameters that represent remifentanil interactions are Theta1 and Theta2, which are unit-less values. Theta1 and Theta2 are zero for all volunteers not receiving remifentanil. In case an interaction between remifentanil and propofol or sevoflurane exists, the estimate for Theta1 will be significantly different from zero. If the interaction in the 4 ng/mL group exceeds the estimated interaction for the 2 ng/mL group, Theta2 will be significantly higher than zero.
Time Frame: 6 weeks
Population: 18 participants experienced the remifentanil 2 ng/mL intervention, and 18 participants experienced the remifentanil 4 ng/mL intervention.
Measure: Mean (Standard Error); unit: Index
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Index
  Theta1, PSI-2 (P): number analyzed (Participants) | 18
  Theta1, PSI-2 (P) | 0 (0)
  Theta1, PSI-2 (S): number analyzed (Participants) | 18
  Theta1, PSI-2 (S) | 0 (0)
  Theta1, PSI-2 (PR 2ng/mL): number analyzed (Participants) | 18
  Theta1, PSI-2 (PR 2ng/mL) | -0.135 (20.8)
  Theta1, PSI-2 (SR 2ng/mL): number analyzed (Participants) | 18
  Theta1, PSI-2 (SR 2ng/mL) | -0.135 (20.8)
  Theta1, PSI-1 (P): number analyzed (Participants) | 18
  Theta1, PSI-1 (P) | 0 (0)
  Theta1, PSI-1 (S): number analyzed (Participants) | 18
  Theta1, PSI-1 (S) | 0 (0)
  Theta1, PSI-1 (PR 2ng/mL): number analyzed (Participants) | 18
  Theta1, PSI-1 (PR 2ng/mL) | -0.135 (20.8)
  Theta1, PSI-1 (SR 2ng/mL): number analyzed (Participants) | 18
  Theta1, PSI-1 (SR 2ng/mL) | -0.135 (20.8)
  Theta2, PSI-2 (P): number analyzed (Participants) | 18
  Theta2, PSI-2 (P) | 0 (0)
  Theta2, PSI-2 (S): number analyzed (Participants) | 18
  Theta2, PSI-2 (S) | 0 (0)
  Theta2, PSI-2 (PR 4ng/mL): number analyzed (Participants) | 18
  Theta2, PSI-2 (PR 4ng/mL) | 0.816 (62.3)
  Theta2, PSI-2 (SR 4ng/mL): number analyzed (Participants) | 18
  Theta2, PSI-2 (SR 4ng/mL) | 0.816 (62.3)
  Theta2, PSI-1 (P): number analyzed (Participants) | 18
  Theta2, PSI-1 (P) | 0 (0)
  Theta2, PSI-1 (S): number analyzed (Participants) | 18
  Theta2, PSI-1 (S) | 0 (0)
  Theta2, PSI-1 (PR 4ng/mL): number analyzed (Participants) | 18
  Theta2, PSI-1 (PR 4ng/mL) | 0.816 (62.3)
  Theta2, PSI-1 (SR 4ng/mL): number analyzed (Participants) | 18
  Theta2, PSI-1 (SR 4ng/mL) | 0.816 (62.3)

ADVERSE EVENTS:
Groups:
- Healthy Volunteers, Propofol (P); Healthy Volunteers, Sevoflurane (S); Healthy Volunteers, Propofol With Remifentanil (PR); Healthy Volunteers, Sevoflurane With Remifentanil (SR): Thirty-six healthy volunteers received four sessions of anesthesia with different common drug combinations while having SedLine EEG sensors placed on their forehead during these sessions to study the effects of these drugs on the brain. The sessions were: propofol (P), sevoflurane (S), propofol with remifentanil (PR), and sevoflurane with remifentanil (SR).
Arm/Group | Healthy Volunteers, Propofol (P) | Healthy Volunteers, Sevoflurane (S) | Healthy Volunteers, Propofol With Remifentanil (PR) | Healthy Volunteers, Sevoflurane With Remifentanil (SR)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 2/36 | 1/36 | 7/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers, Propofol (P) (N=36) | Healthy Volunteers, Sevoflurane (S) (N=36) | Healthy Volunteers, Propofol With Remifentanil (PR) (N=36) | Healthy Volunteers, Sevoflurane With Remifentanil (SR) (N=36)
Vomiting (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain at arterial line site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporary numb sensation in hand (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Short phase of nodale ECG rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days